CLINICAL TRIAL: NCT02293304
Title: Performance of Universal Adhesive in Primary Molars: a Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Rachel de Oliveira Rocha, Rachel de Oliveira Rocha, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TLenzi
Record Dates: First submitted 2014-11-10; First posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-etch approach (Experimental): Application of universal adhesive as self-etch mode
  Interventions: Other: Self-etch approach
- Etch-and-rinse approach (Experimental): Application of universal adhesive as etch-and-rinse mode
  Interventions: Other: Etch-and-rinse approach

INTERVENTIONS:
Other: Self-etch approach — The adhesive will be vigorously agitated on the entire enamel and dentin surfaces for 20 seconds, according to the manufacturer's recommendations.The brush will be scrubbed on the dentin surface under manual pressure followed by gentle air thinning for five seconds and finally light curing for 10 seconds.
  Arms: Self-etch approach
Other: Etch-and-rinse approach — After acid etching for 15 seconds, the sound and caries-affected dentin will be kept moist.The adhesive will be vigorously agitated on the entire enamel and dentin surfaces for 20 seconds, according to the manufacturer's recommendations.The brush will be scrubbed on the dentin surface under manual pressure followed by gentle air thinning for five seconds and finally light curing for 10 seconds.
  Arms: Etch-and-rinse approach

SUMMARY:
The aim of this study is to evaluate the 18-month clinical performance of a multimode adhesive (Scotchbond Universal Adhesive, 3M ESPE, St Paul, MN, USA) in primary molars after partial carious removal. This randomized clinical trial will include subjects (5-10 year-old children) selected at two university centers (UFSM and FOUSP). The sample will consist of 132 primary molars presenting active cavitated carious lesions (with radiographic involvement of the outer half of the dentin), located on the occlusal and occlusal-proximal surface. The sample will be randomly divided into two groups according to bonding approach: etch-and-rinse or self-etch strategy. The restorations will be clinically followed every 6 months for up to 18 months using the USPHS modified criteria for clinical evaluation. Survival estimates for restoration longevity will be evaluated using the Kaplan-Meier method.

DETAILED DESCRIPTION:
Randomized clinical trials of performance of universal adhesive in primary molars

ELIGIBILITY:
Inclusion Criteria:

* active carious lesion in middle dentin limited to the occlusal or occluso-proximal surfaces of primary molars;
* children (male or female) in good general health.

Exclusion Criteria:

* children who refuse or fail to cooperate with the completion of clinical procedure; - teeth without antagonist;
* carious lesions in inner half of dentin;
* presence of painful symptoms or signs of pulpal changes.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Longevity of restoration | 18-month follow up
  The outcome of the study is the failure of restorations in primary teeth. Failures will be assessed by clinical evaluation and will be considered in the presence of loss of restoration or fracture requiring a reintervation (restoration repair or replacement) or symptoms requiring pulp intervention or tooth extraction.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Rocha, Professor, Principal Investigator — Universidade Federal de Santa Maria
Locations (1):
- Federal University of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil